CLINICAL TRIAL: NCT00917527
Title: Randomized Placebo-controlled Crossover Trial of Endothelial Function Improvement in Subjects With History of Premature Coronary Artery Disease
Brief Title: Endothelial Dysfunction in Subjects With History of Premature Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyuk-Jae Chang, Yonsei University, Yonsei University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20090615
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Heart Disease
Keywords: Subjects with family history of coronary heart disease
MeSH Terms: conditions — Coronary Disease | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Atorvastatin
- Atorvastatin (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 40mg/D for 6 weeks to improve endothelial dysfunction

SUMMARY:
The aim of this prospective study is to investigate the prevalence of endothelial dysfunction in subjects with family history of premature coronary heart disease. At the same time, the effect of atorvastatin in treating subclinical endothelial dysfunction in those patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* within 1 year
* the siblings of premature coronary heart disease(male<55years old, female<65years old: Framingham Heart Study)patients admitted relevant hospital

Exclusion Criteria:

* Documented coronary heart disease
* Any woman of childbearing potential who is pregnant, seeking to become pregnant or suspects that she may be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-11 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
improvement of endothelial dysfunction with endo-PAT2000 | 6 weeks later drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Jae Chang, MD, PhD, Principal Investigator — Cardiology Division, Severance Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Nasir K, Michos ED, Rumberger JA, Braunstein JB, Post WS, Budoff MJ, Blumenthal RS. Coronary artery calcification and family history of premature coronary heart disease: sibling history is more strongly associated than parental history. Circulation. 2004 Oct 12;110(15):2150-6. doi: 10.1161/01.CIR.0000144464.11080.14. Epub 2004 Oct 4. PMID 15466626
- [Derived] Hong SJ, Chang HJ, Park S, Kang DR, Shin S, Cho IJ, Shim CY, Hong GR, Ha JW, Chung N. Impact of atorvastatin treatment in first-degree relatives of patients with premature coronary artery disease with endothelial dysfunction: a double-blind, randomized, placebo-controlled crossover trial. Clin Cardiol. 2013 Aug;36(8):480-5. doi: 10.1002/clc.22152. Epub 2013 Jun 10. PMID 23754711